CLINICAL TRIAL: NCT06506968
Title: Quantifying Ergonomic Risk in the Cardiac Catheterization Laboratory: A Comparative Study With and Without a 'Lead-free' Radiation Protection System
Brief Title: Ergonomics in the Cardiac Catheterization Laboratory
Acronym: ERGO-CATH
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Rampart ic, LLC (Unknown)
Responsible Party: Principal Investigator, Ajar Kochar, Program Director for Interventional Cardiology Fellowship, Brigham and Women's Hospital
Other Study IDs: 2023P000484
Record Dates: First submitted 2024-07-10; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Ergonomics; Orthopedic Injury; Wellness
Keywords: Catheterization Laboratory; PCI; CTO; TAVR; Coronary Angiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to quantify ergonomic risk associated with traditional protective equipment in operators working in the cardiac catheterization laboratory as compared with a mobile protection system. The main questions it aims to answer is:

What is the mean time spent by operators in positions of high ergonomic postural risk during cases?

Participants will wear IMU, EMG, and radiation sensors, as well as complete baseline and discomfort surveys for several catheterization procedures.

DETAILED DESCRIPTION:
Study subjects will wear the following equipment on their head and back including: four IMU sensors, eight EMG sensors, and one radiation sensor. Before the catheterization procedure, members of the study team will affix the IMUs on the subject and ensure that the devices are properly calibrated using a calibration procedure as per manufacturer protocol: standing upright with arms and fingers pointing downward and the thumb pointing forward, leaning forward hinging at the hips, and a final pose returning to upright standing position. Participants will periodically be asked to return to upright position to avoid IMU drift. Video of the procedure will also be used for IMU data quality assurance. EMG sensors will also be affixed to the subject and calibrated using the MVC function as per manufacturer protocol: the subject will complete exercises to elicit the maximum muscle activation from each muscle an EMG is placed on. Measures will be taken to reduce EMG impedance including cleaning the skin with alcohol wipes prior to application. One radiation sensor will be clipped to the outside of the participant's clothing, and another will be placed near the left shoulder of the patient as the control.

The IMU sensors will measure body posture angles by the fusion of data from the accelerometer, magnetometer, and gyroscope contained within each sensor. The EMG sensors will measure the muscle activity using non-invasive electrodes on the surface of the skin. The radiation dosimeter will capture radiation received by the participant during each case. The acquired data will be stored locally on the device and upon completion of the procedure, will be removed and the data downloaded by investigator team to the study laptop, offline, utilizing the Ultimum software provided by Noraxon and analyzed with Microsoft Excel and STATA statistical analytic software. Neither the study sponsor RAMPART nor the supplier Noraxon will be permitted to access this data. Specific datasheets will be tabulated per subject and aggregated for time spent in procedures utilizing lead vs procedures in which the RAMPART M1128 device was utilized and lead protective equipment was obviated. Objective EPR will be determined and based on the amount of time the individual body segments were exposed to various postures. Body angles will be assessed and stratified into risk categories (defined as minimal, mild, moderate and high risk and will be assigned modified rapid upper limb risk assessment scores of 1.0, 2.0, 3.0 and 4.0, respectively) and based on the measured body angles in accordance with the modified rapid upper limb assessment During each procedure, the percent time spent in a prespecified range of risk categories for each body part will be calculated. Study staff will mark on a datasheet the procedure type and duration for record. Mean reported discomfort scores will also be calculated at the designated body regions of interest and compared between procedures, as well as with and without the RAMPART device, and across procedure type and duration. Given that the study will be conducted with a single IMU and EMG sensor set, we plan to allow for each subject to utilize the sensor system for up to six cases at a time before rotating to the subsequent subject. This methodology will allow for uninterrupted and less fragmented data acquisition per study subject.

Participants will be asked to complete a baseline survey consisting of questions on demographics, history of orthopedic injury, as well as their years of experience/in practice.

The post procedure surveys will consist of body segment musculoskeletal discomfort ratings.

ELIGIBILITY:
Inclusion Criteria:

* Any member of the BWH cardiac catheterization laboratory who participates in procedures including:
* faculty interventional cardiologists and trainees
* general cardiology fellows
* residents
* physician assistants
* nurses
* circulating and monitoring technologists
* Physically able and willing to wear the sensors required for data collection in the study

Exclusion Criteria:

* Interventionalists not actively participating in the BWH Cardiac Catheterization Lab
* Not able or willing to wear the necessary sensors

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who will be recruited to this study include BWH staff who participate in cardiac catheterization laboratory procedures and consent to be in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mean time spent in positions of high ergonomic risk | May 2024 - December 2024
  This is a directly measurable endpoint utilizing the position and time data acquired from the IMU sensor system and this endpoint will be compared with and without the use of lead protective gear as well as across procedure category and physician reported case complexity. The investigators will report mean time spent in different ergonomic postures stratified by the Rapid Upper Limb Assessment scoring model (1-mild, 2-moderate, 3-high risk, 4-very high risk).

SECONDARY OUTCOMES:
Mean self-reported musculoskeletal discomfort | May 2024 - December 2024
  Participants will report discomfort after each case using a modified cornell muscular discomfort survey. Participants will rate their discomfort from slightly uncomfortable to very uncomfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Ajar Kochar, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No